CLINICAL TRIAL: NCT02969187
Title: Bupivacaine Liposomal Injection (Exparel) for Postsurgical Analgesia in Patients Undergoing Laparoscopic Bariatric Surgery: A Randomized, Double-Blind, Controlled Trial
Brief Title: Bupivacaine Liposomal Injection (Exparel) for Postsurgical Analgesia in Patient Undergoing Laparoscopic Bariatric Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Philip Schauer, Staff Surgeon, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-1318
Record Dates: First submitted 2016-11-09; First posted 2016-11-21 (Estimated); Results first posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Patients at our Bariatric Surgery Center of Excellence fulfilling NIH criteria for bariatric surgery and planned operation of laparoscopic Roux-en Y gastric bypass (LRYGB) or laparoscopic sleeve gastrectomy (LSG) as primary bariatric procedure randomized to receive 20 ml of 1.3% Exparel + 30 ml of 0.5% Bupivacaine + 150 ml of Saline
  Interventions: Drug: Exparel; Drug: Bupivacain; Drug: Saline
- Control (Active Comparator): Patients at our Bariatric Surgery Center of Excellence fulfilling NIH criteria for bariatric surgery and planned operation of laparoscopic Roux-en Y gastric bypass (LRYGB) or laparoscopic sleeve gastrectomy (LSG) as primary bariatric procedure randomized to receive 60ml of 0.5% Bupivacaine + 140 ml of Saline.
  Interventions: Drug: Bupivacain; Drug: Saline

INTERVENTIONS:
Drug: Exparel — 6 trocars are placed to perform LRYGB or LSG: two 12 mm trocars and four 5 mm trocars. Exparel will be injected at port sites.
  Arms: Experimental
Drug: Bupivacain — 6 trocars are placed to perform LRYGB or LSG: two 12 mm trocars and four 5 mm trocars. Bupivacain will be injected at port sites.
Drug: Saline

SUMMARY:
Despite the increasing use of patient-controlled anesthesia (PCA) for postoperative pain management, efforts are continuing to find effective methods to relieve pain after abdominal surgery. Although opioid is an effective analgesic it has opioid related adverse events (ORAEs). Bupivacaine should reduce postoperative pain but it has relatively shorter duration of action. Liposome bupivacaine (Exparel) has been approved as a single dose infiltration for longer postoperative period analgesic. It provides up to 72 hours analgesia postoperatively; results in lesser opioids usage and reduce the ORAEs. Transversus abdominis plane (TAP) block is a relatively new regional anesthetic technique. TAP blocks have been performed to reduce opioid use and control pain in several laparoscopic surgical procedures, including colorectal resections, cholecystectomy and bariatric surgery. The aim of this study is to study the opiate usage, pain and nausea post laparoscopic gastric bypass or sleeve gastrectomy using Exparel versus Bupivacaine as TAP block and port sites infiltration.

DETAILED DESCRIPTION:
Introduction

Despite the increasing use of patient-controlled anesthesia (PCA) for postoperative pain management, efforts are continuing to find effective methods to relieve pain after abdominal surgery. Some studies have already suggested that infusion with local anesthetics at the wound site can decrease postoperative pain levels. Further, other studies have shown equal amounts of opiate analgesic requirements (administered on patient demand) with placebo and local anesthetic administration. However, varying anesthetic administration techniques used in the different studies may explain why the controversy in the literature exists.

Although opioid is an effective analgesic it has opioid related adverse events (ORAEs). Bupivacaine should reduce postoperative pain but it has relatively shorter duration of action. Liposome bupivacaine (Exparel) has been approved as a single dose infiltration for longer postoperative period analgesic. It provides up to 72 hours analgesia postoperatively; results in lesser opioids usage and reduce the ORAEs.

Transversus abdominis plane (TAP) block is a relatively new regional anesthetic technique that targets blockage of the neural afferent of the lower intercostal, iliohypogastric and ilioinguinal nerves in the neurovascular plane between the internal oblique and the transversus abdominis muscle. TAP blocks have been performed to reduce opioid use and control pain in several laparoscopic surgical procedures, including colorectal resections, cholecystectomy and bariatric surgery.

Efficacy of wound infiltration with or without TAP block using immediate-release bupivacaine HCl for acute postsurgical pain is well established; EXPAREL has been proposed as a method for postoperative pain management. Moreover, the administration and the optimal dosage in the bariatric surgical population have not been studied.

The objective of this study is to examine postoperative pain after laparoscopic gastric bypass with TAP block and port sites infiltration using Exparel versus Bupivacaine

Background and significance

Exparel is a FDA approved long-acting, local anesthetic. This is for single-dose infiltration into the surgical site to produce postsurgical analgesia. Exparel offers longer-acting local formulation and can be administered as a single dose. Exparel has a longer duration of action with slower absorption. The mean elimination half-life of local administration of Exparel is approximately 24-34 hours 19-20 versus 2.7 hours for bupivacaine.

Liposomal bupivacaine is for single-dose infiltration and the recommended dose depends on the surgical site but the maximum dose of liposomal bupivacaine is 266 mg and it is injected into soft tissues of the surgical site with frequent aspirations to prevent intravascular injection.

A pooled analysis evaluating the effect of Exparel on pain intensity scores and opioid consumption was published by Dasta et al. This study included 5 surgical procedures (inguinal hernia repair, total knee replacement, hemorrhoidectomy, breast augmentation and bunionectomy) comparing Exparel with bupivacaine HCl, on 912 patients; it showed significantly lower pain score and opioid usage, delayed use of rescue opioid and reduced ORAEs in the Exparel group; as compared to bupivacaine HCL group.

Medication SafetLiposomal bupivacaine has been classified as a high-alert medication by the Institute of Safe Medication Practices due to its similar appearance to propofol. If liposomal bupivacaine were administered intravenously as if it were propofol, adverse cardiac effects may result.

Hypothesis

Exparel (1.3%) and 0.5% Bupivacaine usage with infiltration and TAP block decreases opiate usage, nausea and pain at 48 hours as compared to 0.5% Bupivacaine only.

Primary Objective of the study:

To study the opiate usage, pain and nausea post laparoscopic gastric bypass or sleeve gastrectomy using EXPAREL versus Bupivacaine as TAP block and port sites infiltration.

ELIGIBILITY:
Inclusion Criteria:

* Fulfills NIH criteria for bariatric surgery
* Planned operation of laparoscopic Roux-en Y gastric bypass (LRYGB) or laparoscopic sleeve gastrectomy (LSG) as primary bariatric procedure

Exclusion Criteria:

* BMI <35 and > 60 kg/m2
* Inability to walk (bed-bound or wheelchair dependence)
* Previous major abdominal surgery (possible adhesions and longer operation) defined as:

  * open abdominal surgeries except simple appendectomy and common OB/GYN procedures in the pelvis (hysterectomy, C-section, and oophorectomy, tubal ligation)
  * laparoscopic bowel or solid organ resection except laparoscopic cholecystectomy
  * ventral hernia repair with mesh
* Preoperative chronic opiate use for chronic pain defined as opiate usage at least 60 mg/day of morphine equivalent for ≥ 3 months (as defined by International Association for the Study of Pain22) in the one year period prior to the bariatric surgery
* The American Society of Anesthesiologists (ASA) score > 3
* History of hypersensitivity or adverse reaction to bupivacaine or narcotics
* Inability to speak English
* Concurrent surgical procedure including:

  * ventral hernia repair
  * Cholecystectomy
  * hiatal hernia repair with posterior cruroplasty
  * extensive lysis of adhesions
  * other procedures that mandate addition of "trocar(s)" or "feeding tube"
* Addition of trocar(s) or conversion of surgery to hand-assisted or open

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Patients at our Bariatric Surgery Center of Excellence fulfilling NIH criteria for bariatric surgery and planned operation of laparoscopic Roux-en Y gastric bypass (LRYGB) or laparoscopic sleeve gastrectomy (LSG) as primary bariatric procedure randomized to study arm and control arm.
  6 trocars are placed to perform LRYGB or LSG: two 12 mm trocars and four 5 mm trocars.
  Study arm receive 20 ml of 1.3% Exparel + 30 ml of 0.5% Bupivacaine + 150 ml of Saline (total: 200ml)
  * Transverse Abdominis Plane (TAP) block: 140 ml
  * Port site infiltration:60ml
- Control: Patients at our Bariatric Surgery Center of Excellence fulfilling NIH criteria for bariatric surgery and planned operation of laparoscopic Roux-en Y gastric bypass (LRYGB) or laparoscopic sleeve gastrectomy (LSG) as primary bariatric procedure randomized to study arm and control arm.
  6 trocars are placed to perform LRYGB or LSG: two 12 mm trocars and four 5 mm trocars.
  Control arm receive 60ml of 0.5% Bupivacaine + 140 ml of Saline (total: 200ml)
  * Transverse Abdominis Plane (TAP) block: 140 ml
  * Port site infiltration:60ml
Period: Overall Study
Arm/Group | Experimental | Control
Started | 63 | 63
Completed | 51 | 50
Not Completed | 12 | 13
Not completed — Physician Decision | 12 | 13

BASELINE CHARACTERISTICS:
Population: A total of 101 patients were included; Bupivacaine alone (n=50) and Liposome bupivacaine and bupivacaine (n=51) with a follow up period of 1-month.
Groups:
- Experimental: Patients at our Bariatric Surgery Center of Excellence fulfilling NIH criteria for bariatric surgery and planned operation of laparoscopic Roux-en Y gastric bypass (LRYGB) or laparoscopic sleeve gastrectomy (LSG) as primary bariatric procedure randomized to receive 20 ml of 1.3% Exparel + 30 ml of 0.5% Bupivacaine + 150 ml of Saline
  Exparel: 6 trocars are placed to perform LRYGB or LSG: two 12 mm trocars and four 5 mm trocars. Exparel will be injected at port sites.
  Bupivacain: 6 trocars are placed to perform LRYGB or LSG: two 12 mm trocars and four 5 mm trocars. Bupivacain will be injected at port sites.
  Saline
- Control: Patients at our Bariatric Surgery Center of Excellence fulfilling NIH criteria for bariatric surgery and planned operation of laparoscopic Roux-en Y gastric bypass (LRYGB) or laparoscopic sleeve gastrectomy (LSG) as primary bariatric procedure randomized to receive 60ml of 0.5% Bupivacaine + 140 ml of Saline.
  Bupivacain: 6 trocars are placed to perform LRYGB or LSG: two 12 mm trocars and four 5 mm trocars. Bupivacain will be injected at port sites.
  Saline
- Total: Total of all reporting groups
Arm/Group | Experimental | Control | Total
Number analyzed (Participants) | 51 | 50 | 101
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 41.1 [32.5 to 48.4] | 41.2 [33.7 to 46.8] | 41.1 [32.5 to 48.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 38 | 78
  Male | 11 | 12 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Median (Inter-Quartile Range); unit: kg/m2] — Body mass index
  kg/m2 | 44 [41 to 48] | 44 [42 to 52] | 44 [41 to 48]

OUTCOME MEASURES:

1. Primary Outcome: Total Amount of Opioids at 48 Hours
Description: The total amount of opioids used will be recorded from the nurse chart.
Time Frame: At 48 hours post operative
Population: A total of 126 patients were randomized in this study. Out of that, 25 patients were excluded due either inadequate data, not prescribed post-operative ketorolac or intraoperative additional procedures performed. A total of 101 patients were included;
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Experimental | Control
Number analyzed (Participants) | 51 | 50
mg | 29.5 (17.1) | 27.1 (14.3)

2. Secondary Outcome: Cumulative Pain Score Through 48 Hours After Surgery
Description: Description: We used a time weight average (TWA) pain score in frequent measurements of pain score.
  Cumulative pain score through 48 hours after surgery is the summation of all the time weight average pain scores with a range from 0 to 440.
  The high score represents the worse outcomes. 0 means no pain during the whole time and 440 means severe pain during the whole time.
Time Frame: Pain assessed when the patient is admitted to the recovery room after surgery, every 8 hrs thereafter for up to 48 hours post operatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental | Control
Number analyzed (Participants) | 51 | 50
score on a scale | 177.0 (62.9) | 167.8 (62.3)

3. Secondary Outcome: Cumulative Nausea Score
Description: Description: We used a time weight average (TWA) method in adjusting the nausea score.
  Cumulative nausea score through 72 hours after surgery is the summation of all the time weight average nausea scores with a range from 68-272.
  The high score represents the worse outcomes. 68 means no nausea during the whole time and 272 means severe nausea during the whole time.
Time Frame: Nausea assessed when the patient is admitted to the recovery room after surgery, every 8 hrs thereafter for up to 72 hours post operatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental | Control
Number analyzed (Participants) | 51 | 50
score on a scale | 79 (12) | 98 (35)

ADVERSE EVENTS:
Time Frame: Two patients in the study arm developed urticarial rashes over the abdominal wall at the site of injection. Their rashes were noticed on day 7 after the procedure during follow up visit in the clinic by the attending physician.
Description: Two patients in the study arm developed urticarial rash over the abdominal wall at the site on injection noticed at 1 week post procedure during follow up visit. The rash noticed at 1 week post procedure during follow up visit. The rash was itchy but limited only to the abdominal area at the injection site.
  No other adverse events noted. At subsequent follow up, the rash has resolved.
Arm/Group | Experimental | Control
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/50
Other Adverse Events (participants affected / at risk) | 2/51 | 0/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=51) | Control (N=50)
Minor adverse event (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) — Two patients in the study arm developed urticarial rash over the abdominal wall at the site on injection. The rash was itchy but limited only to the abdominal area at the injection site. At subsequent follow up, the rash has resolved.

LIMITATIONS AND CAVEATS:
There is no data available to guide us on the dosage of liposome bupivacaine in bariatric surgery. We assume adequate quantity and coverage of liposome bupivacaine (266mg) in this obese population, despite that they have a bigger surface area.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-23): https://cdn.clinicaltrials.gov/large-docs/87/NCT02969187/Prot_SAP_000.pdf